CLINICAL TRIAL: NCT06013202
Title: The Efficacy of Nigella Sativa Oil Mouth Rinse in the Management of Recurrent Minor Aphthous Ulcer A Randomized Controlled Clinical Trial With Biochemical Analysis
Brief Title: The Efficacy of Nigella Sativa Oil Mouth Rinse in the Management of Recurrent Minor Aphthous Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nada Sherif (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Nada Sherif, Principal Investiagator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FDASU-RecID032111
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Aphthous Ulcer
Keywords: recurrent; aphthous ulcer; minor; nigella sativa; mouth rinse
MeSH Terms: conditions — Stomatitis, Aphthous; Recurrence | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel randomized control clinical trial
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (TEST GROUP) Nigella Sativa oil mouth rinse (Experimental): Ten patients will receive Nigella Sativa oil mouth rinse. Patients will be asked to use the NS oil mouth rinse (10 ml each 6 hrs.) four times daily . Subjects will be provided with 72 hours supply of the study product. Patients will be instructed to use it for 72 hours with a minimum frequency of four times per day, swished for one minute at each use, in which the first dose was used upon awakening and the last dose just before evening sleep. Patients will be instructed not to use over the counter (OTC) or pharmacy formulated oral rinses or gels during the active treatment phase.
  Interventions: Other: Nigella Sativa Oil Mouth Rinse
- Group 2 (CONTROL GROUP) (Active Comparator): Ten patients will receive the placebo isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl). Patients will be asked to use it as mouth rinse (10 ml each 6 hrs.) four times daily . Subjects will be provided with 72 hours supply of the study product. Patients will be instructed to use it for 72 hours with a minimum frequency of four times per day, swished for one minute at each use, in which the first dose was used upon awakening and the last dose just before evening sleep. Patients will be instructed not to use over the counter (OTC) or pharmacy formulated oral rinses or gels during the active treatment phase.
  Interventions: Other: isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl)

INTERVENTIONS:
Other: Nigella Sativa Oil Mouth Rinse — Nigella Sativa Oil Mouth Rinse
  Arms: Group 1 (TEST GROUP) Nigella Sativa oil mouth rinse
Other: isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl) — isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl)
  Arms: Group 2 (CONTROL GROUP)

SUMMARY:
This research aims to investigate the effectiveness of Nigella Sativa Oil Mouth Rinse application both clinically and biochemically as a suitable affordable treatment modality for Management of Recurrent Minor Aphthous Ulcer

DETAILED DESCRIPTION:
Twenty patients will be selected from the outpatient clinic of the department of Oral Medicine, Periodontology, and Oral diagnosis, Faculty of Dentistry, Ain Shams University and will be divided into two groups (test group and control group), 10 in each group. Ten patients will receive Nigella Sativa oil mouth rinse. Ten patients will receive the placebo isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl). At the screening visit, patient history will be documented, and subjects who met the inclusion/exclusion criteria were asked to complete the survey to determine the severity of their symptoms prior to clinical examination. The oral examination will be a routine visual assessment to document the presence, location and size of an ulcerative oral mucosal lesion.

Patients will be asked to use the NS oil mouth rinse (10 ml each 6 hrs.) four times daily. Subjects will be provided with 72 hours supply of the study product.

Patients will be instructed to use it for 72 hours with a minimum frequency of four times per day, swished for one minute at each use, in which the first dose was used upon awakening and the last dose just before evening sleep. Patients will be instructed not to use over the counter (OTC) or pharmacy formulated oral rinses or gels during the active treatment phase. The same procedure will be done in the control group but by using isotonic (normal saline) with concentration 0.90% of sodium chloride (NaCl). The patients will be re-examined after 24, 48, 72 hrs. from the beginning of the treatment until the complete healing of the (RAU). When patients completed the follow-up phase after product use, they will be asked to repeat the surveys in which they documented the pain scores and oral symptoms. The ulcer size will be measured using periodontal calibrated probe before treatment and after 24, 48, 72 hrs. of treatment until the complete healing of the (RAU).Clinical photographs of the ulcers will be taken using a digital camera preoperatively and after 24, 48, 72 hrs. of treatment until the complete healing of the (RAU). Patients of discomfort and pain severity will be rated at baseline, 24, 48, 72 hours and day seven after using the study product by numeric rating scale (NRS) and visual analog scale for pain (VAS) since, the association between NRS and VAS would be stronger.

The salivary TNF-α levels in RAS patients can be detected by using saliva as a convenient medium and it will be measured prior to the definitive therapy and at the end of using the study product. Distilled water was given to the patients to rinse their oral cavity for 1 minute to remove any debris. Under aseptic conditions, a minimum of 2 ml of saliva will be collected from the patient through 'Spit Technique' after oral rinse with water at room temperature into sterilized tubes every minute for 8-10 minutes. The saliva samples will be collected after one hour or more since the last food intake. The patients will be asked to avoid drinking one hour before sampling. Samples will be immediately frozen at -20°C .The estimation salivary contents of TNF-α will done by enzyme linked immunosorbent assay using a commercial ready-made ELISA kit.

ELIGIBILITY:
Inclusion Criteria:

* All patients should be free from any systemic disease or Behcet syndrome (Atai et al., 2007).
* Patients male or female are eligible (Epstein et al., 2018).
* Oral pain score of 4 or higher on a scale of 0-10 with 0 representing no pain in the presence of oral ulceration (Epstein et al., 2018).
* Patient has only minor aphthous ulcer and its diameter should be less than 1 cm (Atai et al., 2007).
* It should had not been passed more than 4 days from beginning of their ulcer (Atai et al., 2007).

Exclusion Criteria:

* Patients with poor oral hygiene or not willing to perform oral hygiene measures.
* Smoking and alcohol use.
* Pregnant and lactating females.
* Patients with history of any topical or systemic medication or steroid therapy 1 month prior to the investigation (Chaudhuri et al., 2018).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-22 (Estimated); Primary Completion 2024-04-12 (Estimated); Study Completion 2024-09-22 (Estimated)

PRIMARY OUTCOMES:
management of recurrent minor aphthous ulcer as well as patient satisfaction. | 2 week from the baselline
  At the screening visit the discomfort and pain severity of patient's symptoms prior to clinical examination will be rated at baseline, Subjects will be provided with 72 hours supply of the study product. The patients will be re-examined after 24, 48, 72 hrs. and day seven ( a week ) from the beginning of the treatment until the complete healing of the recurrent minor aphthous ulcer which estimated by two week from the baseline. All patients should be with Oral pain score of 4 or higher on a scale of 0-10 with 0 representing no pain in the presence of oral ulceration

SECONDARY OUTCOMES:
Evaluate the effect of Nigella Sativa oil mouth rinse biochemically on the salivary TNF-α level. | 2 week from the baselline
  The salivary TNF-α levels in recurrent minor aphthous ulcer patients will be detected by using saliva as a convenient medium, Salivary samples will be collected at baseline before the intervention and after 24, 48, 72 hrs. and day seven ( a week ) from the beginning of the treatment until the complete healing of the recurrent minor aphthous ulcer which estimated by two week from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nevine Hassan Kheir El Din, Professor, Study Director — Ain Shams University; Ahmed Elsayed Hamed Amr, Lecturer, Study Director — Ain Shams University; Olfat Gameel Shaker, Professor, Study Director — Ain Shams University
Locations (1):
- Nada Mohamed Sherif Aly abdelhamid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No